CLINICAL TRIAL: NCT01466283
Title: Integrative Epigenomic Approach to Gene Discovery in Rhabdomyosarcoma (RMS)
Brief Title: Biomarkers in Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST12B2; COG-ARST12B2 (Other: Children's Oncology Group); ARST12B2 (Other: Children's Oncology Group); NCI-2011-03634 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma
Keywords: childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — DNA Methylation; In Situ Hybridization, Fluorescence; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in patients with rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine genome-wide alterations in DNA methylation in ARMS and ERMS.
* Determine genome-wide DNA copy number alterations in ARMS and ERMS.
* Determine pathogenic genes and pathways by integrative genomic analysis.

OUTLINE: Genome-wide DNA-methylation analysis on ARMS, ERMS, and normal human skeletal myoblasts will be conducted using the HELP (HpaII tiny fragment Enrichment by Ligation-mediated PCR) assay. The methylation status of 1.3 million CpGs at promoters, gene bodies, and intergenic areas will be analyzed. Parallel gene expression analysis will be done and correlated with changes in methylation to uncover genes regulated by epigenetic alterations and altered by genomic losses or gains.

Genes that are altered by both genetic and epigenetic alterations in different sets of patients will be selected by the MIGHT (Multi-dimensional Integration of Genomic data from Human Tissues) algorithm to uncover new genes that are potentially involved in the pathogenesis of ARMS and ERMS. Gene ontology, pathway, and DNA motif analysis algorithms, and other computational approaches will be used to determine the biological consequences of the changes. Prioritized set of epigenetic and genetic alterations will be validated by bisulfite MassArray, FISH, and qRT-PCR in larger numbers of ARMS and ERMS samples.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* 10 ARMS and 10 ERMS frozen samples will be collected from the COG bank via the Cooperative Human Tissue Network (CHTN)
* Human skeletal myoblasts (ZenBio, Research Triangle Park, NC) will serve as controls

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cooperative Human Tissue Network (CHTN)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Genome-wide alterations in DNA methylation in ARMS and ERMS
Genome-wide DNA copy number alterations in ARMS and ERMS
Pathogenic genes and pathways by integrative genomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Y. Hu, MD, Principal Investigator — Tomorrows Children's Institute at Hackensack University Medical Center